CLINICAL TRIAL: NCT07149701
Title: Ventricular Tachycardia Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025135
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Ventricular Tachycardia (VT)
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal treatment: Treatment without intervention of catheter ablation or Implantable cardioverter defibrillator.
  Interventions: Device: Intervention

INTERVENTIONS:
Device: Intervention — Treatment with intervention of catheter ablation or Implantable cardioverter defibrillator.

SUMMARY:
The goal of this observational study is to detect the long-term risk of a composite endpoint event in adult patients with ventricular tachycardia (VT) who are managed with catheter ablation or non-ablation management (including modern drug therapy and/or ICD therapy).

ELIGIBILITY:
Inclusion Criteria:

* Sustained ventricular tachycardia (VT), defined as VT lasting ≥30 seconds or requiring intervention due to hemodynamic compromise within 30 seconds; or Clinically significant non-sustained VT (NSVT) where the treating clinician has determined that therapeutic intervention is necessary.

Exclusion Criteria:

* Concurrent participation in any interventional clinical trial that, in the judgment of the investigator, could interfere with the data collection or outcome assessment of this observational study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with ventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite of death and recurrence of ventricular tachycardia | 1 year

IPD SHARING:
Plan to Share IPD: Undecided